CLINICAL TRIAL: NCT03235401
Title: "Validation of a Questionnaire Assessing Disability and Bothersomeness in Pulmonary Arterial Hypertension (PAH): The PAH Disability and Bothersomeness Questionnaire"
Brief Title: The PAH Disability and Bothersomeness Questionnaire
Acronym: PAH-DBoQ
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Association de Recherche en Physiopathologie Respiratoire (Other)
Collaborators: GlaxoSmithKline (Industry); Soladis (Industry); Interlis (Unknown)
Responsible Party: Sponsor
Other Study IDs: PAH-DBoQ
Record Dates: First submitted 2017-07-28; First posted 2017-08-01 (Actual); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Pulmonary Arterial Hypertension (PAH)
Keywords: Questionnaire; Disability assessment; Bothersomeness; Pulmonary Arterial Hypertension; patient-reported outcome measure; New York Heart Association (NYHA) functional class
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pulmonary Arterial Hypertension patients
  Interventions: Other: 37-items questionnaire

INTERVENTIONS:
Other: 37-items questionnaire — Patient will answer the PAH-DBoQ questionnaire

SUMMARY:
To develop a patient-reported questionnaire to investigate the impact of PAH (pulmonary arterial hypertension) on patients' daily lives in terms of bothersomeness and disability.

DETAILED DESCRIPTION:
A 3-steps study protocol was initiated in 2011 to develop a patient reported outcome measure (PROM) in PAH.The first two steps have been completed (qualitative study and Delphi consensus study) leading to the development of a provisional 37-items questionnaire. A reduction of items in this provisional questionnaire and the validation of the final questionnaire are the goals of the current study.

ELIGIBILITY:
Inclusion Criteria:

* patients with idiopathic and heritable PAH;
* patients over 18;
* male and female;
* NYHA Functional Class I, II, III & IV;
* Written consent signed
* Patients with a good understanding of the French - language
* Patient affiliated with a social security scheme

Exclusion Criteria:

* Patients under 18 years of age
* Patients with other pathologies associated with PAH (Group 1)
* Patients with other forms of pulmonary hypertension (groups 2, 3, 4 and 5)
* Non-consenting patients
* Patients who do not have a good understanding of the French language

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: * 120 patients with idiopathic and heritable PAH (40 of which will be selected for a test-retest procedure)
  * Patients with PAH associated with other diseases will be excluded in order to clearly circumscribe the results to PAH
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2017-06-16 (Actual); Primary Completion 2017-12-16 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
Cronbach's alpha≥ 0.7 | at the end of the study (an average of 6 months)
  Internal consistency of the PAH Disability and Bothersomeness Questionnaire will be assessed with Cronhbach's alpha

SECONDARY OUTCOMES:
Low rate of answers (≤95%) | at the end of the study (an average of 6 months)
  low rate of answers will help reducing the number of questionnaire's items

CONTACTS AND LOCATIONS:
Overall Officials: Olivier SITBON, PHD, Principal Investigator — Service de Pneumologie et Soins Intensifs, Hôpital de Bicêtre, Université Paris-Sud France
Locations (1):
- Centre de Référence de l'Hypertension Pulmonaire Sévère, Service de Pneumologie et Soins Intensifs, Hôpital de Bicêtre,, Le Kremlin-Bicêtre, Val De Marne, France

IPD SHARING:
Plan to Share IPD: No